CLINICAL TRIAL: NCT01574898
Title: Pilot Pharmacokinetic Study of Three New Nicotine Lozenge Formulations (V0474) Versus Two Reference Formulations (V0018 B mg and Niquitin® Fresh Mint, 4mg) After Single Oral Administration in Healthy Male Smokers.
Brief Title: Pilot Pharmacokinetic Study of New Nicotine Lozenge Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V00474 PC 1 01; 2012-000419-94 (EudraCT Number)
Record Dates: First submitted 2012-04-02; First posted 2012-04-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Smokers
Keywords: Smoking cessation; Nicotine; Tobacco Use Disorder; Central Nervous System Agents
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

ARMS (5):
- Niquitin® Fresh Mint 4 mg (Active Comparator)
  Interventions: Drug: Niquitin® Fresh Mint 4 mg
- V0118 - B mg (Active Comparator)
  Interventions: Drug: V0018 - B mg
- V0474 - C mg (Experimental)
  Interventions: Drug: V0474 - C mg
- V0474 - B mg (Experimental)
  Interventions: Drug: V0474 - B mg
- V0474 - A mg (Experimental)
  Interventions: Drug: V0474 - A mg

INTERVENTIONS:
Drug: V0474 - A mg — Single oral administration
  Arms: V0474 - A mg
Drug: V0474 - B mg — Single oral administration
  Arms: V0474 - B mg
Drug: V0474 - C mg — Single oral administration
  Arms: V0474 - C mg
Drug: V0018 - B mg — Single oral administration
  Arms: V0118 - B mg
Drug: Niquitin® Fresh Mint 4 mg — Single oral administration
  Arms: Niquitin® Fresh Mint 4 mg

SUMMARY:
The purpose of this study is to determine the pharmacokinetic profile of nicotine following a single oral administration of three new nicotine lozenge formulations (V0474) in comparison with two reference products. The clinical and biological safety of V0474 and the lozenge acceptability will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject aged 18 to 45 years (inclusive)
* Current smoker of < or = 10 cigarettes/day
* Fagerström score < or = 5
* Absence of any clinically significant abnormal finding at physical, ECG, biological examinations in the Investigator's opinion

Exclusion Criteria:

* Presence of any significant medical finding or significant history (in particular any cardio-vascular disease, severe renal or hepatic insufficiency, current gastric or duodenal ulcer or oesophagitis) that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator
* Current or recurrent buccal lesions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of nicotine following a single oral nicotine lozenge administration in healthy smokers | 12 time points up to 6h after oral administration
  Pharmacokinetic profile of nicotine following a single oral nicotine lozenge administration in healthy smokers by measuring Maximum Plasma Concentration (Cmax), Time of Maximum Concentration (Tmax) , Area under the nicotine plasma concentration curve (AUC0-t), for each test and reference formulations

SECONDARY OUTCOMES:
Clinical safety (reported adverse events) | Screening up to Day 5
  Safety by evaluating the number of subjects with emergent adverse events and changes from baseline to end of study in vital signs, Electrocardiogram (ECG) and clinical laboratory parameters.
Acceptability questionnaire | Up to complete lozenge dissolution, about 30 minutes (4 times)
  Quantitative and qualitative descriptive analysis of the scores reported by treatment and assessment time

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France